CLINICAL TRIAL: NCT01869257
Title: Impact of Triclosan-coated Suture on Surgical Site Infection After Colorectal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Luca Vittorio Gianotti, Researcher, University of Milano Bicocca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-SSI 09; UNIMIB18 (Other: Milano-Bicocca University)
Record Dates: First submitted 2013-05-24; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Resection
Keywords: triclosan; colorectal; surgery; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator): regular suture not coated with triclosan
  Interventions: Device: regular suture
- triclosan (Experimental): Experimental group will receive abdominal wound closure with suture matherial that is coated with triclosan
  Interventions: Device: Triclosan coated suture

INTERVENTIONS:
Device: Triclosan coated suture — The patients in the treated arm will have the abdominal wound sutured with triclosan-coated suture
  Arms: triclosan
Device: regular suture — The control arm will have the abdominal wound sutured with a regular non-coated suture
  Arms: control

SUMMARY:
Despite adequate antimicrobial prophylaxis and perioperative correction of risk factors, surgical site infections (SSI) remain the most frequent complication of colorectal resection (range 10-17%). Several strategies may be implemented to prevent SSI. Among these, the use of local antimicrobial agents seems successful.

The primary aim of the present trial was to evaluate the efficacy of a surgical suture, coated with Triclosan a synthetic soluble antimicrobial agent, in reducing the SSI rate after colorectal operations.

DETAILED DESCRIPTION:
This was a non-sponsored, multicenter, prospective, randomized, controlled, single-blind study. Two hundred and seventy-three patients candidate to colorectal resection were enrolled. Exclusion criteria were: age < 18 or > 85 years, pregnancy, peritonitis, peritoneal contamination during operation, ongoing infections, ASA score > 3, denied consent.

135 were randomized to the treatment arm and 136 to the control arm. Treatment consisted of abdominal wound closure by suturing peritoneum, fascia, subcutaneous tissue, and skin with Polyglactin 910 Triclosan-coated suture (treatment arm) or with Polyglactin without Triclosan (control arm). SSI were defined according to the Atlanta CDC. Patients were followed up by office visits for 30 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients candidate to elective colorectal resection

Exclusion Criteria:

* no consent
* peritonitis
* hypersensitivity to triclosan
* ASA > 3
* ongoing infections

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2009-05; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Rate of surgical site infection | 30 days
  the incidence of superficial and deep wound infection in patients who underwent colorectal resection will be determined by a blind observer according to the Atlanta CDC definition.
  The unit of measure will be number of wound infection over the number of treated or control patients

SECONDARY OUTCOMES:
overall wound complications | 30 days

OTHER OUTCOMES:
length of hospital stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Nespoli, MD, Study Chair — Milano-Bicocca University
Locations (1):
- San Gerardo Hospital, Monza, Italy

REFERENCES:
- [Background] Chang WK, Srinivasa S, Morton R, Hill AG. Triclosan-impregnated sutures to decrease surgical site infections: systematic review and meta-analysis of randomized trials. Ann Surg. 2012 May;255(5):854-9. doi: 10.1097/SLA.0b013e31824e7005. PMID 22470067
- See also: Related Info — http://www.ncbi.nlm.nih.gov/